CLINICAL TRIAL: NCT02343718
Title: A Study of Vinblastine and Temsirolimus in Pediatric Patients With Recurrent or Refractory Lymphoma or Solid Tumours Including CNS Tumours
Brief Title: Vinblastine and Temsirolimus in Pediatrics With Recurrent or Refractory Lymphoma or Solid Tumours Including CNS Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I218
Record Dates: First submitted 2015-01-13; First posted 2015-01-22 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Recurrent Lymphoma; Refractory Lymphoma; Solid Tumours; Central Nervous System
MeSH Terms: conditions — Lymphoma | interventions — Vinblastine; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vinblastine and Temsirolimus (Experimental): Vinblastine starting dose:
  Weight >12 kg 4mg/m^2 Weight ≤ 12 kg 0.13mg/kg IV push for 1 minute Days 1, 8, 15, 22, 29 and 36. Cycle length is 6 weeks up to 6 cycles.
  Temsirolimus starting dose:
  Weight >12 kg 15mg/m^2 Weight ≤ 12 kg 0.5 mg/kg IV for 1 hour on days 1, 8, 15, 22, 29 and 36. Cycle length is 6 weeks up to 6 cycles.
  Interventions: Drug: Vinblastine; Drug: Temsirolimus

INTERVENTIONS:
Drug: Vinblastine
Drug: Temsirolimus

SUMMARY:
The purpose of this study is to determine the best dose of vinblastine that can be given with a new drug, temsirolimus.

DETAILED DESCRIPTION:
Vinblastine is already approved in the treatment of some types of cancer in children and temsirolimus is already used to treat some adult cancers in Canada. Temsirolimus has been shown to slow the growth of tumours in animals but it is not known if it can also slow tumour growth in children. Laboratory studies suggest that giving both vinblastine and temsirolimus may offer better results than giving vinblastine alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological verification of malignancy at initial diagnosis or at relapse.

Note: Histological verification is not required for patients with optic pathway gliomas, or patients with pineal tumours and elevations of CSF or serum tumour markers

* Solid tumours (excluding soft tissue sarcomas), CNS and localized brainstem tumours (excluding diffuse intrinsic pontine gliomas (DIPG)) or,
* Lymphomas including Hodgkin's disease, non-Hodgkin's lymphoma and post-transplant lymphoproliferative disease (PTLD)
* Patients must have relapsed or refractory disease for which there is no known curative therapy, with either measurable or evaluable disease
* Age ≥ 1 year and ≤ 18 years at time of registration
* Performance status:

  * Patients ≤ 16 years: Lansky ≥ 50%
  * Patients ≥ 16 years: Karnofsky > 50%

Prior Therapy

Patients must have received at least one prior regimen prior to registration. There is no limit to the number of prior regimens. Patients must have recovered from the acute effects and reversible toxicities related to prior therapy and have adequate washout prior to study entry as follows:

Surgery:

Previous major surgery is permitted provided that it has been at least 28 days prior to registration and wound healing has occurred. Additionally, at least 7 days must have elapsed since last biopsy or other minor surgery and wound healing must have occurred.

Radiation:

Prior radiotherapy is permitted provided that from last dose to registration:

* At least 90 days have elapsed from total body irradiation, craniospinal radiotherapy or if ≥ 50% radiation of pelvis.
* At least 6 weeks have elapsed from other substantial bone marrow irradiation.
* At least 2 weeks have elapsed from local palliative radiotherapy (small port),
* At least 8 weeks have elapsed from 131I-MIBG therapy for neuroblastoma.

Chemotherapy:

Prior myelosuppressive chemotherapy is permitted provided that it has been at least 3 weeks (6 weeks if nitrosurea) from last administration.

Prior therapy with vinblastine, mTOR inhibitors (such as temsirolimus or sirolimus) is permitted provided patients did not develop progressive disease during treatment and patients have never had to discontinue treatment due to severe adverse events such as interstitial lung disease. At least 3 weeks must have elapsed from the last administration of these agents and registration.

Other Therapy:

Patients may have received other therapies provided that an adequate time has elapsed from completion of therapy/last dose as follows:

* At least 60 days from stem cell transplant/rescue without total body irradiation and no signs of graft-versus-host disease (GVHD).
* At least 7 days (2 weeks for peg-filgrastim) from completion of therapy with hematopoietic growth factors.
* At least 3 half-lives from last administration of monoclonal antibodies.
* At least 6 weeks from any other immunotherapy (e.g. vaccines).
* For biologic anti-neoplastic agents, the longer of the following must have elapsed from last administration prior to study entry: At least 2 weeks or, Standard cycle length of prior regimen or, 5 half-lives.

  - Adequate Bone Marrow Function, defined as:
* Absolute neutrophil count (ANC) ≥ 1.0x10^9/L.
* Platelets ≥ 100 x 10^9/L (transfusion independent defined as not receiving platelet transfusions within 7 days prior to registration).
* Hemoglobin > 80 g/L (may receive RBC transfusions). Patients with known bone marrow disease will be eligible for the study provided they meet bone marrow criteria above and they are not known to be refractory to red cell or platelet transfusions.

  - Adequate Renal Function, defined as:
* Measured creatinine clearance/GFR ≥ 70 mL/min/1.73 m2 OR,
* Serum creatinine ≤ 1.5 x ULN for age.

  - Adequate Liver Function, defined as:
* Total bilirubin ≤ 1.5 x upper limit normal for age.
* ALT ≤ 1.5 x upper limit of normal.
* Serum albumin ≥ 20 g/L.

  - Adequate Metabolic Function, defined as:
* Serum triglyceride level ≤ 3.42 mmol/L (300 mg/dL).
* Serum cholesterol level ≤ 7.75 mmol/L (300 mg/dL).
* Blood glucose ≤ ULN for age. Initial sampling may be random; if abnormal, fasting blood glucose must be obtained and be within the upper normal limits for age.
* Adequate Pulmonary Function, defined as:

  * No dyspnea at rest.
  * O2 saturations of ≥ 92% on room air.
  * Patients with any baseline respiratory symptoms, or with a history of pulmonary toxicity, and who are old enough to complete pulmonary function tests, should have documented FEV1 and vital capacity ≥ 50% normal value.
* Electrolytes: ≤ grade 1 (Potassium, Calcium, Magnesium, Phosphate)
* Patient or guardian consent must be obtained on all patients according to local Institutional and/or University Human Experimentation Committee requirements. Children > 8 years old whose parent or guardian has signed consent on their behalf may also sign assent if desired
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient registration

Exclusion Criteria:

* Patients with serious illness or medical condition that would not permit the patient to be managed according to the protocol including, but not limited to:

  1. Active or uncontrolled infections;
  2. Uncontrolled diabetes;
  3. Any other medical conditions that might be aggravated by treatment;
  4. History of an underlying inherited or ongoing bleeding disorder;
  5. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events (e.g. heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age) or mean resting corrected QT interval (QTc) > 470 msec).
* Patients with a history of allergic reactions or known hypersensitivity to the study drug(s) or their components, or compounds of similar chemical or biologic composition.
* Patients with lymphoma or solid tumours (except primary CNS tumours) who have untreated brain metastases, untreated spinal cord compression or meningeal metastases are not eligible (CNS imaging is not required to rule this out unless there is a clinical suspicion of CNS disease). Patients with treated brain metastases who have radiologic evidence of stable brain metastases, with no evidence of cavitation or hemorrhage in the brain lesion, are eligible providing that they are asymptomatic. If being treated with corticosteroids, must be at a stable or decreasing dose for at least 7 days prior to study entry.
* Concurrent Medications

  * Patients receiving other investigational agents.
  * Patients receiving other anti-cancer agents, or radiation therapy.
  * Patients receiving angiotensin-converting enzyme (ACE) inhibitors.
  * Patients receiving QT/QTc-prolonging drugs.
  * Patients receiving anticoagulants.
  * Patients receiving anti-GVHD or agents to prevent organ rejection post-transplant.
  * Patients receiving strong/potent CYP3A4/5 substrates/inhibitors/inducers. These agents must have been discontinued for at least 14 days prior to registration. Grapefruit juice is also not permitted for at least 14 days prior to registration and at any time during study participation.
* Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use a highly effective contraceptive method. Pregnant or breast feeding females will not be entered on this study due to the potential fetal and teratogenic adverse events.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 4 years
  To determine the recommended phase II dose (RP2D) of the combination of vinblastine and temsirolimus (administered as a weekly intravenous dose) in children with recurrent or refractory solid tumours including central nervous system (CNS) tumours and lymphoma and to describe the associated toxicities in children

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Baruchel, Study Chair — Hospital for Sick Children, Toronto ON Canada; Rebecca Deyell, Study Chair — Children's & Women's Health Centre of BC Branch, Vancouver BC, Canada
Locations (6):
- Canada (6):
  - Children's and Women's Health Centre of BC Branch, Vancouver, British Columbia
  - Izaak Walton Killam (IWK) Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deyell RJ, Wu B, Rassekh SR, Tu D, Samson Y, Fleming A, Bouffet E, Sun X, Powers J, Seymour L, Baruchel S, Morgenstern DA. Phase I study of vinblastine and temsirolimus in pediatric patients with recurrent or refractory solid tumors: Canadian Cancer Trials Group Study IND.218. Pediatr Blood Cancer. 2019 Mar;66(3):e27540. doi: 10.1002/pbc.27540. Epub 2018 Nov 4. PMID 30393943